CLINICAL TRIAL: NCT04916574
Title: Clinical Trial of Nasal Spray Containing Anti-SARS-CoV-2 Antibodies Derived From Bovine Colostrum
Brief Title: Clinical Trial of BioBlock COVID-19 Nasal Spray Containing Anti-SARS-CoV-2 Antibodies Derived From Bovine Colostrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icosagen Cell Factory (Industry)
Collaborators: Tartu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ico-CT001
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: SARS-COV2 Infection; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioBlock® concentration 0.2 mg/mL (Active Comparator): BioBlock®: Nasal Spray Containing Anti-SARS-CoV-2 Antibodies Derived from Bovine Colostrum
  Interventions: Other: Nasal Spray Containing Anti-SARS-CoV-2 Antibodies Derived from Bovine Colostrum
- BioBlock® concentration 0.1 mg/mL (Active Comparator): BioBlock®: Nasal Spray Containing Anti-SARS-CoV-2 Antibodies Derived from Bovine Colostrum
  Interventions: Other: Nasal Spray Containing Anti-SARS-CoV-2 Antibodies Derived from Bovine Colostrum

INTERVENTIONS:
Other: Nasal Spray Containing Anti-SARS-CoV-2 Antibodies Derived from Bovine Colostrum — Concentration of active substance on nasal mucosal surface in time

SUMMARY:
For an antiviral agent to act as an effective biological barrier on nasal mucosal surface, the formulation preferably has to be maintained on the site of action for several hours, and the nasal spray dispenser can be utilized for administering the solution to the upper respiratory tract. A "first-in-man" clinical study of the nasal spray containing anti-SARS-CoV-2 antibodies derived from bovine colostrum was conducted. The study on healthy volunteers was undertaken to evaluate how long the bovine antibodies would be maintained on the nasopharyngeal surface after administration of nasal spray. In addition, the study enabled to determine which of the two concentrations of antibodies should be used in the final nasal-spray formulation. The volunteers were followed up for 4h after administration of antibody spray and sampling was done at different time-points during this period. The concentration of antibodies from patient samples was measured using ELISA analysis. In addition, as this was a "first-in-man" study any adverse events following the administration of spray were also monitored.

DETAILED DESCRIPTION:
To test the nasal biological availability of the BioBlock® immunoglobulin preparation, 16 healthy volunteers were recruited in the phase 0 clinical trial. The study was conducted in the premises of the Ear Clinic of Tartu University Hospital. The study protocol was approved by Research Ethics Committee of the University of Tartu on March 17, 2021 (No 336/T-1). Written informed consent in accordance with the Declaration of Helsinki was obtained from each healthy volunteer. The study group was divided into two subgroups where the individuals were intranasally administered into both nostrils of BioBlock® formulation which contained either 0.1 mg/mL or 0.2 mg/mL of the colostrum immunoglobulin preparation (n=8 in both study groups). A filter paper with a volume capacity of 15 µL was placed on the medial nasal surface using surgical forceps and it was kept on nasal mucosa for 10 minutes. Following this the BioBlock was administered to the nasal cavity. The nasal mucosal sampling was done at 4 timepoints. The samples were analyzed using a Cow IgG ELISA kit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Age 18-80
* Have not been diagnosed with SARS-COV-2 infection (lack of positive PCR test)
* Have not been vaccinated against SARS-COV-2 infection

Exclusion Criteria:

* Pregnancy
* Serious allergic or anaphylactic reactions to medications
* Allergies to milk products
* Ear-nose-throat pathologies (anatomic and diseases)
* Immunodeficiency conditions (cancers, hematologic diseases, HIV, congenital immunodeficiency)
* Viral hepatitis A,B and C
* Upper airway infections
* Autoimmune diseases (diabetes, COPD, asthma, rhinitis, RA, psoriasis)
* Concomitant drugs - glucocorticosteroids, biologic drugs, inhalable medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Antibody concentration dynamics | 4 hours
  Concentration of bovine IgG at different timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Icosagen AS, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Undecided